CLINICAL TRIAL: NCT06031181
Title: Sublobar Resection for Adenocarcinoma in Situ/Minimally Invasive Adenocarcinoma Diagnosed by Intraoperative Frozen Section: a Single-arm, Multi-center, Phase III Trial
Brief Title: Sublobar Resection for Adenocarcinoma in Situ/Minimally Invasive Adenocarcinoma Diagnosed by Intraoperative Frozen Section (ECTOP-1019)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Haiquan Chen, Director in the Department of Thoracic Surgery, FUSCC, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SAFROS
Record Dates: First submitted 2023-09-04; First posted 2023-09-11 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Lung Adenocarcinoma; Frozen Section; Sublobar Resection
MeSH Terms: conditions — Adenocarcinoma of Lung

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sublobar resection (Experimental): Sublobar resection is performed for Adenocarcinoma in Situ/Minimally Invasive Adenocarcinoma Diagnosed by Intraoperative Frozen Section
  Interventions: Procedure: Sublobar Resection

INTERVENTIONS:
Procedure: Sublobar Resection — Sublobar Resection includes segmentectomy and wedge resection

SUMMARY:
This is a clinical trial from Eastern Cooperative Thoracic Oncology Project (ECTOP), numbered as ECTOP-1019. The goal of this clinical trial is to confirm the therapeutic effect of sublobar resection for AIS/MIA diagnosed by intraoperative frozen section.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who sign the informed consent form and are willing to complete the study according to the plan;
2. Aged from 18 to 80 years old;
3. ECOG equals 0 or 1;
4. Not receiving lung cancer surgery before;
5. Resectable peripheral cT1N0M0 tumors;
6. Single lung nodules with ground-glass dominant or pure ground-glass on CT, or multiple lung nodules with the major lesion being the aforementioned nodules;
7. Adenocarcinoma in Situ/Minimally Invasive Adenocarcinoma Diagnosed by Intraoperative Frozen Section
8. Not receiving chemotherapy or radiotherapy before.

Exclusion Criteria:

1. Not cT1N0M0;
2. Cannot be completely resected by sublobar resection;
3. Invasive lung adenocarcinoma or not lung adenocarcinoma diagnosed cytologically or pathologically;
4. Receiving lung cancer surgery before;
5. Receiving radiotherapy or chemotherapy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 390 (Estimated)
Dates: Start 2023-03-31 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
5-year recurrence-free survival | 5 years
  The event is defined as the tumor recurrence.

SECONDARY OUTCOMES:
5-year overall survival | 5 years
  The event is defined as the death due to any causes.

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zheng S, Deng C, Li Y, Zhang Y, Chen H. Sublobar resection for adenocarcinoma in situ and minimally invasive adenocarcinoma diagnosed by intraoperative frozen section (ECTOP-1019): a study protocol of prospective, single-arm, multicenter, phase III study. J Thorac Dis. 2024 Sep 30;16(9):6286-6291. doi: 10.21037/jtd-24-623. Epub 2024 Sep 18. PMID 39444881